CLINICAL TRIAL: NCT00379496
Title: A Randomized Controlled Trial of Acupuncture Added to Usual Treatment for Fibromyalgia
Brief Title: Trial of Acupuncture Added to Usual Treatment for Fibromyalgia
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of Sao Paulo (Other)
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 843/99
Record Dates: First submitted 2006-09-21; First posted 2006-09-22 (Estimated); Last update posted 2006-09-22 (Estimated); Status verified 2006-09

CONDITIONS: Fibromyalgia
Keywords: Fibromyalgia; Acupuncture; Randomized study
MeSH Terms: conditions — Fibromyalgia | interventions — Antidepressive Agents; Acupuncture Therapy

INTERVENTIONS:
Procedure: Antidepressants
Procedure: acupuncture

SUMMARY:
The aim of this study was to evaluate the effect of acupuncture as a treatment for this condition. Fifty-eight women diagnosed with fibromyalgia were randomly allocated to two groups. One group received acupuncture (n=34) twice a week for 20 sessions in addition to tricyclic antidepressants and exercises. The control group (n=24) received only tricyclic antidepressants and exercises. A blinded assessor evaluated patients' pain using visual analog scale (VAS), tender points number (TePsN) and myalgic index (MI). The same assessor also evaluated quality of life (QoL) using SF-36. These evaluations were done prior to treatments, at the end of the 20 sessions, and again at six months, one year and two years after the first evaluation. At the end of the 20 sessions, patients who had received acupuncture were significantly better than those who had not in all measures of pain (VAS, TePsN, MI) and in five subscales of SF-36. After six months, the acupuncture group was significantly better than the control group in some measures of pain (TePsN and MI) and in three subscales of SF-36. After one year, the acupuncture group showed significant advantage in only one subscale of SF-36; at two years there were no significant differences between the two groups on all outcome measures. The addition of acupuncture to usual treatment for fibromyalgia is beneficial for pain and quality of life, but only in first six months.

DETAILED DESCRIPTION:
Fibromyalgia is a diffuse musculoskeletal pain syndrome with multiple tender points which are widely and symmetrically distributed throughout the body. The main symptom is widespread musculoskeletal pain, lasting longer than three months, which is associated with chronic fatigue, cognitive dysfunction, sleep disorder, morning stiffness, anxiety and depression. The etiology of fibromyalgia remains unknown.

In Brazil, fibromyalgia is estimated to affect two-and-half percent of the population . This incidence is similar to other countries .Acupuncture, which involves inserting needles at specific points on the patient's skin, is one of the oldest forms of therapy and is widely practiced in the United States. Each year about one million Americans undergo acupuncture treatments, mainly to relieve pain caused by a variety of ailments . A consensus statement from the U.S. National Institutes of Health (NIH) concluded that acupuncture may be useful as an adjunct treatment or may be an acceptable alternative treatment in a comprehensive management program for fibromyalgia patients (NIH Consensus Conference, 1998.In Brazil, there is increased interest in acupuncture; in 1995, a federal law established that the procedure can only be performed by physicians.

Systematic reviews looking at the effectiveness of acupuncture for fibromyalgia have found a limited amount of high quality scientific studies. These reviews concluded that acupuncture was more effective than sham (placebo) acupuncture in improving symptoms of fibromyalgia. There is a need for acupuncture trials that include a large sample size of patients with similar and well-defined pain conditions. Such trials should utilize standardized and well-described acupuncture stimuli. These should be placed effectively in the skin in accordance with classical Chinese experience and utilizing unequivocal primary outcome measures for the effect.

ELIGIBILITY:
Inclusion Criteria:

* Patients had to report moderate to severe pain intensity (VAS > four), and they had to be using antidepressant medication in an analgesic dose (between 12.5mg/day and 75mg/day).

Exclusion Criteria:

* Patients were excluded in the case of severe psychiatric disease, the presence of neurological deficits, cardiac disease or glaucoma, and treatment with acupuncture within one year prior to the start of the study.

Ages: 20 Years to 70 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 58
Dates: Start 2000-04; Study Completion 2002-05

PRIMARY OUTCOMES:
VAS(Visual Analogical Scale)
SF-36(Short Form 36)
Myalgic Index
Number of tender points

SECONDARY OUTCOMES:
VAS(Visual Analogical Scale)(5 times)
SF-36(Short Form 36)(5 times)
Myalgic Index(5 times)
Number of tender points(5 times)

CONTACTS AND LOCATIONS:
Overall Officials: Rosa A Targino, MD, Principal Investigator — University of Sao Paulo-School of Medicine
Locations (1):
- Hospital das Clinicas da Faculdade de Medicina da Universidade de Sao Paulo, São Paulo, São Paulo, Brazil